CLINICAL TRIAL: NCT05436717
Title: Efficacy and Implementation of an Online Mindfulness and Compassion-based Program (MINDxYOU) for Reducing Stress and Promote Mental Health Among Healthcare Providers in Spain
Brief Title: Efficacy and Implementation of MINDxYOU Program for Reducing Stress and Promote Mental Health Among Healthcare Providers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Miguel Servet (Other)
Responsible Party: Principal Investigator, Javier Garcia Campayo, Principal Investigator, Hospital Miguel Servet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI22/341
Record Dates: First submitted 2022-06-22; First posted 2022-06-29 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Mental Health Wellness
Keywords: Healthcare providers; Stress; Third-wave psychotherapies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MINDxYOU (Experimental): The online program MINDxYOU is based on the principles of 'third wave' psychotherapies, such as the promotion of wellbeing through the practice of mindfulness, compassion, acceptance, and spirituality and the estimated time for completing the whole program is 8 weeks
  Interventions: Behavioral: MINDxYOU

INTERVENTIONS:
Behavioral: MINDxYOU — The online program MINDxYOU is based on the principles of 'third wave' psychotherapies and it is an online program particularly addressed at healthcare providers which will both monitor and support the individual's mental health. The program is self-administered and will be delivered via the Internet and available via smartphone, tablet, and personal computer.

SUMMARY:
Because of the COVID-19 pandemic situation, social and health professionals constitute a population in risk of developing psychopathologies due to the high levels of stress they experience. There is consensus regarding the need of offering these professionals psychotherapeutic evidence-based interventions addressed to reducing their stress levels and promote their wellbeing; because of the current situation, it is believed that online interventions might be the best-fitted approach. The research groups that present this project have leaded a research line that has proved the efficacy of online psychotherapeutic programs in the past. In the present project, the efficacy of the MINDxYOU program will be evaluated; this is an online intervention based on mindfulness techniques, compassion, and acceptance, and that has been developed specifically for social and health professionals. In addition, in order to overcome the gap that separates the validation of interventions and their posterior implementation, this project aims to perform an implementation study in which a hybrid design will be adopted to test the impact of the program in terms of efficacy and the feasibility of the implementation. The investigators will adopt the framework proposed by Hermes. et al., inspired in Proctor's recommendations. The study will be conducted in 2 autonomous communities (Aragón and Andalucía).

ELIGIBILITY:
Inclusion Criteria:

* Working as a doctor, nurse, physiotherapist, psychologist, nursing assistant, ambulance technician, or being a trainee student in any health profession, or working in a nursing home.
* Aged between 18 and 70.
* Ability to understand Spanish.
* Digital literacy and access to a smartphone, tablet, or personal computer with Internet connection.
* Giving informed consent.

Exclusion Criteria:

* Presenting an illness that affects the central nervous system.
* Having a diagnosis of a severe psychiatric condition (including severe depressive disorders, suicidal tendencies, bipolar disorders, panic disorders, anxiety or stress-related disorders, obsessive-compulsive disorders, and substance-related disorders).
* Presenting a medical, infectious, or degenerative illness that is not under control.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS) | Baseline
  Consists of 10 items in which participants are asked to rate how unpredictable, uncontrollable, and overloaded they have found their life over the past month on a 5-point Likert-type scale. Scores range from 0 to 40, and higher scores reflect higher levels of perceived stress.
Perceived Stress Scale (PSS) | Post-treatment 10 weeks from baseline
  Consists of 10 items in which participants are asked to rate how unpredictable, uncontrollable, and overloaded they have found their life over the past month on a 5-point Likert-type scale. Scores range from 0 to 40, and higher scores reflect higher levels of perceived stress.
Perceived Stress Scale (PSS) | 6 months follow-up from baseline
  Consists of 10 items in which participants are asked to rate how unpredictable, uncontrollable, and overloaded they have found their life over the past month on a 5-point Likert-type scale. Scores range from 0 to 40, and higher scores reflect higher levels of perceived stress.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Baseline
  It is a 9-item scale aimed at screening for depression in primary care and other medical settings. It assesses the frequency of depressive symptoms during the last 2 weeks using a scale from 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 27, with higher scores indicating higher severity of depression.
Patient Health Questionnaire (PHQ-9) | Post-treatment 10 weeks from baseline
  It is a 9-item scale aimed at screening for depression in primary care and other medical settings. It assesses the frequency of depressive symptoms during the last 2 weeks using a scale from 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 27, with higher scores indicating higher severity of depression.
Patient Health Questionnaire (PHQ-9) | 6 months follow-up from baseline
  It is a 9-item scale aimed at screening for depression in primary care and other medical settings. It assesses the frequency of depressive symptoms during the last 2 weeks using a scale from 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 27, with higher scores indicating higher severity of depression.
General Anxiety Disorder-7 (GAD-7) | Baseline
  It is a 7-item self-reported measure to assess the intensity of anxiety symptoms. It refers to the period of the past 2 weeks; each item is scored in a 4-point Likert-type scale, resulting in a total score that can range from 0 to 21, with higher values reflecting more severe anxiety symptoms.
General Anxiety Disorder-7 (GAD-7) | Post-treatment 10 weeks from baseline
  It is a 7-item self-reported measure to assess the intensity of anxiety symptoms. It refers to the period of the past 2 weeks; each item is scored in a 4-point Likert-type scale, resulting in a total score that can range from 0 to 21, with higher values reflecting more severe anxiety symptoms.
General Anxiety Disorder-7 (GAD-7) | 6 months follow-up from baseline
  It is a 7-item self-reported measure to assess the intensity of anxiety symptoms. It refers to the period of the past 2 weeks; each item is scored in a 4-point Likert-type scale, resulting in a total score that can range from 0 to 21, with higher values reflecting more severe anxiety symptoms.
Brief Symptoms Inventory (BSI) | Baseline
  It is a 18-item self-reported questionnaire designed to offer a rapid screening of symptoms of psychological disorders. Each item is scored in a 5-point Likert-type scale, reflecting on the past 7 days.
Brief Symptoms Inventory (BSI) | Post-treatment 10 weeks from baseline
  It is a 18-item self-reported questionnaire designed to offer a rapid screening of symptoms of psychological disorders. Each item is scored in a 5-point Likert-type scale, reflecting on the past 7 days.
Brief Symptoms Inventory (BSI) | 6 months follow-up from baseline
  It is a 18-item self-reported questionnaire designed to offer a rapid screening of symptoms of psychological disorders. Each item is scored in a 5-point Likert-type scale, reflecting on the past 7 days.
Connor-Davidson Resilience Scale (CD-RISC) | Baseline
  It is a 10-item self-reported measure addressed at assessing resilience. Each item is scored in a 5-point Likert scale, and the total score, which ranges from 1 to 5, is calculated by averaging the scores of the items; higher scores indicate higher levels of resilience.
Connor-Davidson Resilience Scale (CD-RISC) | Post-treatment 10 weeks from baseline
  It is a 10-item self-reported measure addressed at assessing resilience. Each item is scored in a 5-point Likert scale, and the total score, which ranges from 1 to 5, is calculated by averaging the scores of the items; higher scores indicate higher levels of resilience.
Connor-Davidson Resilience Scale (CD-RISC) | 6 months follow-up from baseline
  It is a 10-item self-reported measure addressed at assessing resilience. Each item is scored in a 5-point Likert scale, and the total score, which ranges from 1 to 5, is calculated by averaging the scores of the items; higher scores indicate higher levels of resilience.
Five Facets of Mindfulness Questionnaire -15 item version (FFMQ-15) | Baseline
  It is an adaptation of the original 39-item FFMQ, a questionnaire addressed at measuring the five facets of mindfulness. Each subscale of the FFMQ-15 includes 3 items, scored in a Likert-type scale (1-5). A score for each subscale, ranging from 5 to 15, can be computed by summing the items, where higher scores indicate higher levels of the mindfulness facet.
Five Facets of Mindfulness Questionnaire -15 item version (FFMQ-15) | Post-treatment 10 weeks from baseline
  It is an adaptation of the original 39-item FFMQ, a questionnaire addressed at measuring the five facets of mindfulness. Each subscale of the FFMQ-15 includes 3 items, scored in a Likert-type scale (1-5). A score for each subscale, ranging from 5 to 15, can be computed by summing the items, where higher scores indicate higher levels of the mindfulness facet.
Five Facets of Mindfulness Questionnaire -15 item version (FFMQ-15) | 6 months follow-up from baseline
  It is an adaptation of the original 39-item FFMQ, a questionnaire addressed at measuring the five facets of mindfulness. Each subscale of the FFMQ-15 includes 3 items, scored in a Likert-type scale (1-5). A score for each subscale, ranging from 5 to 15, can be computed by summing the items, where higher scores indicate higher levels of the mindfulness facet.
Sussex-Oxford Compassion Scales (SOCS) | Baseline
  This scale is composed by two 20-item self-report scales measuring compassion. A total score, ranging from 20 to 100, is calculated for each scale, and higher total values indicate higher levels of compassion
Sussex-Oxford Compassion Scales (SOCS) | Post-treatment 10 weeks from baseline
  This scale is composed by two 20-item self-report scales measuring compassion. A total score, ranging from 20 to 100, is calculated for each scale, and higher total values indicate higher levels of compassion
Sussex-Oxford Compassion Scales (SOCS) | 6 months follow-up from baseline
  This scale is composed by two 20-item self-report scales measuring compassion. A total score, ranging from 20 to 100, is calculated for each scale, and higher total values indicate higher levels of compassion
Acceptance and Action Questionnaire-II (AAQ-II) | Baseline
  It is a measure for assessing experiential avoidance, a key element of 'third wave' psychotherapies that refers to the tendency to avoid thoughts, feelings, memories, sensations and other internal experiences, and which is very commonly associated with worse mental health outcomes, as opposite to psychological flexibility. The scale presents 7 items scored in a 7-point Likert-type scale, and a total score is calculated by summing all the items. Higher scores mean higher experiential avoidance.
Acceptance and Action Questionnaire-II (AAQ-II) | Post-treatment 10 weeks from baseline
  It is a measure for assessing experiential avoidance, a key element of 'third wave' psychotherapies that refers to the tendency to avoid thoughts, feelings, memories, sensations and other internal experiences, and which is very commonly associated with worse mental health outcomes, as opposite to psychological flexibility. The scale presents 7 items scored in a 7-point Likert-type scale, and a total score is calculated by summing all the items. Higher scores mean higher experiential avoidance.
Acceptance and Action Questionnaire-II (AAQ-II) | 6 months follow-up from baseline
  It is a measure for assessing experiential avoidance, a key element of 'third wave' psychotherapies that refers to the tendency to avoid thoughts, feelings, memories, sensations and other internal experiences, and which is very commonly associated with worse mental health outcomes, as opposite to psychological flexibility. The scale presents 7 items scored in a 7-point Likert-type scale, and a total score is calculated by summing all the items. Higher scores mean higher experiential avoidance.
EuroQol five-dimensional classification system (EQ-5D) | Baseline
  It is a widely used health-related quality of life measure. First, the participant is asked to report how severe (1= no problems, 2= mild, 3= moderate, 4= severe, 5= extreme) are the problems they may present in the day of reporting regarding each of the following five domains: mobility, self-care, usual activities, pain, and anxiety/depression. The utility scores are obtained from the EQ-5D classification system and are used to rate patients' health-related quality of life, which normally range from 0 (although it is possible to present negative scores) to 1 (i.e., "perfect health").
EuroQol five-dimensional classification system (EQ-5D) | 6 months follow-up from baseline
  It is a widely used health-related quality of life measure. First, the participant is asked to report how severe (1= no problems, 2= mild, 3= moderate, 4= severe, 5= extreme) are the problems they may present in the day of reporting regarding each of the following five domains: mobility, self-care, usual activities, pain, and anxiety/depression. The utility scores are obtained from the EQ-5D classification system and are used to rate patients' health-related quality of life, which normally range from 0 (although it is possible to present negative scores) to 1 (i.e., "perfect health").
Client Service Receipt Inventory (CSRI) | Baseline
  It is addressed at describe and measure service utilization patterns as a basis for estimating associated costs across healthcare, social care and community settings.
Client Service Receipt Inventory (CSRI) | 6 months follow-up from baseline
  It is addressed at describe and measure service utilization patterns as a basis for estimating associated costs across healthcare, social care and community settings.
System Usability Scale (SUS) | Post-treatment 10 weeks from baseline
  It is a 10-item questionnaire to measure the usability which qualitatively is related with the quality and acceptability of the intervention. The scale presents 5-point Likert-type scale (0 = never, 1 = almost never, 2 = often, 3 = sometimes and 4 = always). A total score, ranging from 0 to 40, is calculated by totalling the scores from all the items, and higher total values indicate higher level of acceptability of the intervention
Client Satisfaction Questionnaire adapted to Internet-Based interventions (CSQ-I) | Post-treatment 10 weeks from baseline
  It is an 8-item, 4-point Likert scale questionnaire that assesses the general satisfaction of the participants regarding the received intervention. The total score ranges from 8 to 32.
Intervention Appropriateness Measure (IAM) | Post-treatment 10 weeks from baseline
  Includes 4 items designed to measure appropriateness of the intervention. The scale presents 5-point Likert-type scale (1 = completely disagree, 2 = in disagreement, 3 = neither agree nor disagree, 4 = agree and 5 = completely agree). A total score, ranging from 0 to 20, is calculated by totalling the scores from all the items, and higher total values indicate higher level of appropriateness of the intervention
Attitudes towards Psychological Online Interventions (APOI) | Post-treatment 10 weeks from baseline
  Includes 16 items to assess attitudes toward online interventions among people with depressive symptomatology. The APOI explores four dimensions; "Skepticism and Perception of Risks", "Confidence in Effectiveness", "Technologization Threat" and "Anonymity Benefits". Each factor is calculated from the sum of 4 specific items. The scale presents 5-point Likert-type scale (1 = totally agree, 2 = agree, 3 = I'm not sure, 4 = disagree and 5 = totally disagree). Each factor can get a score between 4-20 points, and the higher the score, the greater the sensation perceived by the participant in each of the factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry. Miguel Servet University Hospital, Zaragoza, Spain

REFERENCES:
- [Derived] Lopez-Del-Hoyo Y, Fernandez-Martinez S, Perez-Aranda A, Monreal-Bartolome A, Barcelo-Soler A, Camarero-Grados L, Armas-Landaeta C, Guzman-Parra J, Carbonell V, Campos D, Chen X, Garcia-Campayo J. Effectiveness of a Web-Based Self-Guided Intervention (MINDxYOU) for Reducing Stress and Promoting Mental Health Among Health Professionals: Results From a Stepped-Wedge Cluster Randomized Trial. J Med Internet Res. 2025 Feb 3;27:e59653. doi: 10.2196/59653. PMID 39899345
- [Derived] Lopez-Del-Hoyo Y, Fernandez-Martinez S, Perez-Aranda A, Barcelo-Soler A, Guzman-Parra J, Varela-Moreno E, Campos D, Monreal-Bartolome A, Beltran-Ruiz M, Moreno-Kustner B, Mayoral-Cleries F, Garcia-Campayo J. Effectiveness and implementation of an online intervention (MINDxYOU) for reducing stress and promote mental health among healthcare workers in Spain: a study protocol for a stepped-wedge cluster randomized trial. BMC Nurs. 2022 Nov 10;21(1):308. doi: 10.1186/s12912-022-01089-5. PMID 36357881